CLINICAL TRIAL: NCT02882568
Title: Analysis of Immune Response In Bacterial Infection of Obese Subject
Acronym: ARIIBO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Roderick Meckenstock, Dr, Versailles Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: P15/19_ARIIBO
Record Dates: First submitted 2016-06-14; First posted 2016-08-30 (Estimated); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- investigational (Other): Blood test for Inflammatory and immunological analysis during acute sepsis phase and one month later
  Interventions: Biological: blood analysis

INTERVENTIONS:
Biological: blood analysis — Pilot study, single center, interventional including 15 obese subjects with acute sepsis. Inflammatory and immunological tests during acute phase and one month later after a presumed return parameters at baseline

SUMMARY:
Improve knowledge of the immune response to sepsis in obese patients. Define immunological and genetic prognostic factors of severe infections which can motivate a change in the therapeutic attitude

ELIGIBILITY:
Inclusion Criteria:

* between18 and 80 years
* obesity: BMI > 30
* presumed bacterial infection:

  * pneumonitis (documented or probably)
  * pyelonephritis / acute prostatitis
  * soft tissue / skin infection (except for bedsore)
  * cholecystitis / angiocholitis
  * meningitis
  * clostridium colitis
  * surgical site infection
* signed consent

Exclusion Criteria:

* patients with viral, parasitic or mycotic documented infection
* patients with bacterial infection with treatment> 4 weeks (ex. endocarditis; osteo- articular infections)
* patients with prior antibiotic treatment (< 14 days)
* intensive care unit patients
* patients with a history of cancer or malignant hematological disease within the 5 previous years that is currently clinically significant (non metastatic prostatic and basocellular malignancy are excluded)
* patients with systemic disease
* Known diagnosis of human immunodeficiency infection (DICV, HIV…)
* immunosuppression treatment during last month including corticotherapy
* pregnancy
* 3 months follow up not possible
* non signed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-08; Primary Completion 2016-02 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Patterns of inflammatory and immunological markers in obese patients in sepsis and post- sepsis ("normal") situation | T 0 and at 1 month
  Standard inflammatory markers; immunological markers (cytokines, leptine, lymphocyte phenotype)

SECONDARY OUTCOMES:
Evaluation of sepsis; correlation with inflammatory and immunological parameters | T 0 and at 1 month
Analysis of leptine polymorphism | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Ch de Versailles, Le Chesnay, France